CLINICAL TRIAL: NCT03552419
Title: A Multidisciplinary Approach to Peripartum Triaging of Patients to the Operating Room: A Quality Improvement Project
Brief Title: A Quality Improvement Project - Peripartum Operating Room Leveling System
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00164177
Record Dates: First submitted 2018-05-02; First posted 2018-06-11 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2020-08

CONDITIONS: Pregnancy Complications; Cesarean Section Complications; Morbidity;Perinatal
Keywords: Operating room leveling; Obstetric anesthesia; Time to incision
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Level Red: A level red refers to a case with an immediate threat to the life of the fetus or mother and may not be delayed under any circumstance.
- Level Orange: A level orange case requires the patient to arrive in the OR within 30 minutes from the time of decision with the approximate estimated time of arrival determined by the obstetrician.
- Level Yellow: A level yellow case requires operative intervention, but there is no maternal and/or fetal compromise at the time of evaluation. Timing to the OR is agreed upon by both the anesthesiology and obstetrical providers. The case may be delayed if a level red or orange case is identified. Possible
- Level Green: A level green case is most dependent on the acuity of the OR suite and unit. The patient and/or fetus are stable with no threat to the health of either.

SUMMARY:
Investigators propose a four-category triaging system to delineate and facilitate the communication and action plan for all types of obstetric OR cases via a multidisciplinary approach. Investigators omitted ambiguous terms and developed an algorithm to categorize patients according to acuity and risk. Investigators' quality improvement intervention allows for rapidly changing circumstances and accounts for both obstetric and anesthetic considerations.

Several metrics will be collected to evaluate this multidisciplinary quality improvement project, including maternal demographics, labor characteristics, and indication for surgical intervention. Additional data include level assigned, time of patient arrival in OR, type of surgery performed, and anesthetic delivered. Investigators will collect fetal delivery data, including Apgar scores and umbilical cord gases, as well as maternal delivery data, including estimated blood loss, time to uterine incision and delivery, and surgical complications.

DETAILED DESCRIPTION:
At investigators' institution, a triage (or leveling) system for emergency surgeries in the general operating rooms (OR) exists with the goal of optimizing patient care and reducing morbidity and mortality. In the obstetric field, while medical terminology exists for these situations to delineate and convey the urgency of a particular peripartum situation, for example "stat, emergent, or urgent," it is generally acknowledged that this terminology is not universal and is somewhat ambiguous, causing confusion and unnecessary delays in patient care.

Investigators propose a quality improvement project which will delineate terminology for obstetrical triaging to the OR and discuss metrics for evaluation of this quality improvement intervention. Investigators developed a multidisciplinary stratification system at investigators' institution to triage obstetric patients into a four-level system with clear guidelines for all OR cases. Investigators' categorization system accounted for maternal and fetal stability, indication for surgical intervention, role for obtaining additional studies, nil per os (NPO) status, and surgical and anesthetic concerns. Within each of the four classifications, investigators defined the expectations for each team member's role, including the obstetrician, anesthesiologist, charge nurse, nursing staff, neonatal intensive care unit (NICU) team, and the surgical and clinical technicians.

Several metrics will be collected to evaluate this multidisciplinary quality improvement project, including maternal demographics, labor characteristics, and indication for surgical intervention. Additional data include level assigned, time of patient arrival in OR, type of surgery performed, and anesthetic delivered. Investigators will collect fetal delivery data, including Apgar scores and umbilical cord gases, as well as maternal delivery data, including estimated blood loss, time to uterine incision and delivery, and surgical complications.

ELIGIBILITY:
Inclusion Criteria:

* Female of child-bearing age, requiring emergent procedure in operating room (including cesarean section, D&C, cerclage placement or removal)

Exclusion Criteria:

* Patients not requiring urgent surgical or invasive procedures

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female of child-bearing age
Study Population: In obstetrics, triage assessment incorporates both maternal and fetal considerations. Priority is given to situations with obvious threat to life to the mother or to the fetus. While medical terminology exists for these situations to delineate and convey the urgency of a particular peripartum situation, for example "stat, emergent, or urgent," it is generally acknowledged that this terminology is not universal and is somewhat ambiguous, causing confusion and unnecessary delays in patient care. Furthermore, simply classifying the need for cesarean into a single "emergency" category is insufficient as varying levels of "emergencies" exist. In the modern-day era, the obstetrical decision for surgical intervention prompts the mobilization of a team of providers, including the obstetrician, anesthesiologist, nursing and surgical technicians, and supporting OR staff. Thus, effective communication among team members is essential.
Sampling Method: Non-Probability Sample
Enrollment: 1380 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Materno-fetal stability | 1 year
  This will be assessed by ICU admissions (days) and total length of hospital stay (days)
Indication for surgical intervention | 1 year
  surgery is required if patient has one or more of the following reasons: non-reassuring fetal tracing, umbilical cord prolapse, peripartum hemorrhage, or emergency dilation and curettage.
Role for obtaining additional studies | 1 year
  determine by the number of additional testing including Labs, imaging or EKG a patient required on top of standard studies.
nil per os (NPO) status | 1 year
  Time of last intake (fluid or solids) measured in hours and minutes
Surgical concerns | 1 year
  Concerns that may change our care, i.e. patient is full stomach but needs to have urgent surgery. This will be assessed via observation of patient condition and need of hospital care

CONTACTS AND LOCATIONS:
Overall Officials: Jamie D Murphy, MD, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No